CLINICAL TRIAL: NCT06879353
Title: Comparison of Efficacy of Single Dose Tranexamic Acid Versus Placebo Before Surgery in Females Undergoing Surgery for Ovarian Cancer
Brief Title: Comparison of Single-Dose Tranexamic Acid Vs. Placebo in Ovarian Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Kainat usman, Principal Investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheikh ZMC/H1
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; Perioperative Blood Loss; Blood Transfusion Events
Keywords: Ovarian Neoplasms; Tranexamic Acid; Perioperative Blood Loss; Gynecologic Oncology
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Tranexamic Acid (Experimental): Participants in this group received a single preoperative intravenous dose of tranexamic acid at 15 mg/kg before undergoing surgery for ovarian cancer.
  Interventions: Drug: Tranexamic Acid (TXA)
- Group Placebo (Placebo Comparator): Participants in this group received an equal volume of normal saline as a placebo intravenously before undergoing surgery for ovarian cancer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — A single intravenous dose of tranexamic acid (15 mg/kg) was administered before surgery to assess its efficacy in reducing perioperative blood loss and the need for transfusion.
  Arms: Group Tranexamic Acid
Drug: Placebo — An equal volume of intravenous normal saline was administered as a placebo before surgery to compare outcomes with the tranexamic acid group.
  Arms: Group Placebo

SUMMARY:
This study evaluated the effectiveness of a single dose of tranexamic acid compared to a placebo in reducing blood loss and the need for blood transfusions in women undergoing surgery for ovarian cancer. Tranexamic acid, a medication that helps control bleeding by stabilizing blood clots, has been widely used in other surgical settings but has not been well studied in ovarian cancer surgery.

Participants were randomly assigned to receive either a single dose of tranexamic acid or a placebo before surgery. Blood loss was measured during and after the procedure, and the need for blood transfusions was recorded. The study aimed to determine whether tranexamic acid was effective in reducing perioperative blood loss and minimizing the need for transfusions.

The findings contributed to understanding whether this cost-effective and widely available medication could improve surgical outcomes and reduce complications associated with excessive bleeding in ovarian cancer patients.

DETAILED DESCRIPTION:
After obtaining approval from the ethical committee and CPSP and securing informed consent from the participants, all females who met the inclusion criteria were enrolled in the study from the outpatient department of OBGYN, Sheikh Zayed Medical College, Rahim Yar Khan. Their ASA status was assessed by a consultant anesthesiologist and documented by the researcher, along with their FIGO stage of cancer, which was determined by a consultant radiologist with a minimum of two years of experience. Patient demographics, including age, weight (measured by the researcher using a weighing scale), height (measured by the researcher using a wall-mounted height scale in meters), BMI (in kg/m²), duration of ovarian cancer, menstrual status (menstruating/menopausal), history of chemotherapy exposure, and prior abdomino-pelvic surgery (assessed by reviewing previous surgical records), were recorded.

Patients were then randomly divided into two groups using the paper lottery method:

Group (A) - Tranexamic Acid Group received a single preoperative dose of intravenous tranexamic acid at 15 mg/kg.

Group (B) - Placebo Group received an equal volume of normal saline. Patients were blinded to their group assignments. The surgery was performed by a consultant surgeon with at least three years of experience. Perioperative blood loss was calculated by the researcher as per the operational definition. Patients with post-operative hemoglobin levels below 9 g/dL, assessed through a CBC report obtained within 12 hours after surgery, were transfused with packed red blood cells.

Efficacy was assessed based on the requirement for transfusion after surgery, and it was labeled positive if no transfusion was needed. All data were documented using a self-designed proforma. Patient anonymity and confidentiality were maintained as a priority, with no personal identifiers such as patient names or contact details included in the documentation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60.
* Female gender.
* Ovarian cancer of > 12 months duration.
* FIGO stage I-III.
* American Society of Anesthesiologists (ASA) status 1-3.

Exclusion Criteria:

1. Ovarian cancer of FIGO stage IV
2. ASA status 4-6.
3. Hypersensitivity to tranexamic acid, (assessed by reviewing previous medical record).
4. History of bleeding or clotting disorders (assessed by reviewing previous medical record).
5. Impaired renal function (serum creatinine > 1.3 mg/dl).
6. History of coronary heart disease (assessed by reviewing previous medical record).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only Females
Enrollment: 372 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Requirement of Blood Transfusion After Surgery | Within 12 hours after surgery
  The proportion of patients requiring a blood transfusion after surgery due to post-operative hemoglobin levels falling below 9 g/dL. Efficacy was defined as the absence of transfusion requirement postoperatively.

SECONDARY OUTCOMES:
Perioperative Blood Loss | During surgery and within 12 hours postoperatively
  Perioperative blood loss was calculated using the formula:
  Perioperative Total Blood Loss (mL) = 1000 × (Preoperative Hemoglobin - Postoperative Hemoglobin) / Preoperative Hemoglobin The measurement provided an objective assessment of blood loss during and immediately after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kainat Usman, Principal Investigator — Sheikh Zayed Medical college/Hospital, Rahimyar Khan
Locations (1):
- Sheikh Zayed Medical college/hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No